CLINICAL TRIAL: NCT06196918
Title: Efficacy and Safety of Rivaroxaban in the Prevention of Venous Thromboembolism in Glioma Patients With Postoperative Lower Extremity Dyskinesia
Brief Title: Efficacy and Safety of Rivaroxaban in the Prevention of Venous Thromboembolism in Glioma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NFEC-2023-314
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Glioma, Malignant
Keywords: Glioma; Rivaroxaban; Venous Thromboembolism; Dyskinesia
MeSH Terms: conditions — Glioma; Venous Thromboembolism; Dyskinesias | interventions — Rivaroxaban; Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban group (Experimental): Patients with highly suspected, newly diagnosed, untreated glioma undergo surgical resection. CT scan within 24 hours after surgery is performed to rule out intracranial hemorrhage and/or infarction. Then those patients with postoperative lower extremity dyskinesia are treated with rivaroxaban (10 mg/day) and compression stockings until 1 month after surgery.
  Interventions: Drug: Rivaroxaban 10 MG
- Placebo group (Active Comparator): Patients with highly suspected, newly diagnosed, untreated glioma undergo surgical resection. CT scan within 24 hours after surgery is performed to rule out intracranial hemorrhage and/or infarction. Then those patients with postoperative lower extremity dyskinesia are treated with placebo and compression stockings until 1 month after surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rivaroxaban 10 MG — Patients with postoperative lower extremity dyskinesia are treated with rivaroxaban (10 mg/day) and compression stockings until 1 month after surgery.
  Other Names: Jiangsu Zhongbang pharmaceutical CO., LTD; Serial numbers: H20203733
  Arms: Rivaroxaban group
Drug: Placebo — Patients with postoperative lower extremity dyskinesia are treated with placebo (10 mg/day) and compression stockings until 1 month after surgery.
  Other Names: Jiangsu Zhongbang pharmaceutical CO., LTD
  Arms: Placebo group

SUMMARY:
Glioma is a common brain tumor with a high risk of venous thromboembolism during treatment, especially in the months after surgery. Postoperative lower extremity dyskinesia in patients with gliomas is considered as a high-risk factor for venous thromboembolism. Rivaroxaban, as an oral anticoagulants, has similar effect in the prevention and treatment of tumor-related venous thromboembolism compared to low molecular weight heparin. Given the lack of prospective supporting data, the efficacy and safety of rivaroxaban in the prevention of postoperative venous thromboembolism in glioma patients with postoperative lower extremity dyskinesia need to be established.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is a disorder in which blood clots abnormally in the veins, resulting in complete or incomplete blockage of blood vessels, including deep vein thrombosis and pulmonary embolism of the lower extremities, and is a common complication in patients with malignancy. In a retrospective analysis of the causes of death in patients with active cancer receiving chemotherapy, thromboembolic disease was the second leading cause of death, with VTE accounting for the vast majority. The risk of venous thromboembolism varies depending on the type of cancer, but it has been reported that the incidence of brain tumors can be greater than 20 percent per year, especially in the early postoperative period. High-grade gliomas are common brain tumors with a 20 to 30 percent risk of venous thrombosis during treatment, and postoperative lower extremity dysfunction in patients with high-grade gliomas is considered a high-risk factor for venous thrombosis. Because many high-grade gliomas are located in or adjacent to functional areas, such as frontopariparietal glioma, parietal glioma, thalamic glioma, and others, patients are more likely to develop limb dysfunction. Therefore, it is necessary to prevent venous thromboembolism for patients with high-grade glioma with lower extremity dysfunction after surgery.

Risk factors for venous thromboembolism can be divided into patient-related, tumor-related, and treatment-related. Patient-related factors include age >65 years, weight gain, hypertension, A or AB blood type, previous history of venous thrombosis or pulmonary embolism, and paraparesis. Risk factors associated with tumors include high-grade glioma, tumor diameter >5 cm, and residual tumor after surgery. Treatment-related risk factors include early postoperative period (within 30 days), surgery time >4 hours, chemotherapy, anti-vascular endothelial growth factor therapy, hormonal therapy, and central venous catheterization. Lower extremity dysfunction in patients with glioma is both tumor-related and treatment-related. In the past, clinicians did not routinely administer prophylactic anticoagulation to glioma patients with lower limb disorders because the use of anticoagulants would increase the chance of postoperative intracranial hemorrhage. However, it was reported that the risk of venous thromboembolism in patients with lower extremity dysfunction was 2.6 to 3.6 times than in those without lower extremity dysfunction, and recent studies have shown that the combination of perioperative compression stockings, pneumatic plantar venous pumps and low molecular weight heparin (LMWH) maximizes the prevention of venous thromboembolism in critically neurosurgical patients without a high risk of bleeding. Moreover, a previous randomized, double-blind prospective clinical trial evaluated the safety of heparin in the perioperative period of brain tumors, and the results suggested that the perioperative use of low-dose heparin in brain tumors was safe and effective, and did not increase the risk of bleeding compared with controls. Another meta-analysis further confirmed the safety of LMWH or unfractionated heparin for the prevention of venous thromboembolism after neurosurgery.

However, there are few studies on the use of LMWH in this population, and there is no consensus on the safety of LMWH for the prevention of venous thromboembolism in this population. A phase III randomized controlled trial in patients with high-grade glioma, initiated in 2002, evaluated the safety and efficacy of postoperative LMWH for the prevention of venous thromboembolism, suggesting that LMWH can reduce the occurrence of venous thrombosis but also increase the risk of bleeding. The Eastern Cooperative Oncology Group has also evaluated the use of LMWH for the prevention of glioblastoma, and the use of LMWH reduced thrombosis without increasing the probability of intracranial hemorrhage. In addition, the scale and number of cases in the above studies were small. Therefore, there is an urgent need to explore an effective and safe method to prevent postoperative venous thromboembolism in glioma patients with lower limb dysfunction.

Rivaroxaban is an oral anticoagulant that directly inhibits Xa and thrombin and is widely used in noncancer-associated VTE due to its oral availability, high bioavailability with no need for frequent coagulation monitoring. In the study of tumor-related VTE, rivaroxaban has preliminarily shown no less effect than LMWH in the prevention and treatment of venous thromboembolism. Mohamed et al. systematically reviewed and meta-analyzed the efficacy and complications of LMWH and rivaroxaban in cancer-related thrombosis, and the results suggested that rivaroxaban had a lower risk of VTE recurrence and all-cause mortality, and that the main bleeding risk was no different from that of LMWH. In a phase III SELECT-D pilot study comparing the efficacy and complications of cancer-related thrombosis with the two agents, rivaroxaban was associated with a low risk of VTE recurrence and a low risk of major and non-major bleeding. Therefore, rivaroxaban has a good role in the prevention of tumor-related VTE. And because of its convenience of being oral and not requiring frequent monitoring, it is of great significance for clinical treatment.

In summary, in view of the current lack of research on postoperative prophylactic anticoagulation therapy in patients with glioma, our center plans to lead a multi-center, randomized, double-blind controlled prospective clinical trial in glioma patients with lower limb dysfunction after surgery. To determine whether the addition of rivaroxaban has a more active preventive effect on postoperative venous thromboembolism, and to explore the safety of rivaroxaban in preventing postoperative venous thromboembolism in glioma patients lower limb dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-80 years old with highly suspected (as assessed by study surgeon), newly diagnosed, untreated glioma.
* Patients without heart insufficiency, lungs insufficiency, renal insufficiency, hepatic insufficiency, autoimmune diseases and other organ diseases with severe dysfunction.
* Individuals who agree to undergo surgical resection.
* Individuals with dyskinesia after surgery.
* All patients giving written informed consent.

Exclusion Criteria:

* Individuals with age < 18 years or > 80 years.
* Patients with heart insufficiency, lungs insufficiency, renal insufficiency, hepatic insufficiency, autoimmune diseases and other organ diseases with severe dysfunction.
* Individuals have acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhea), have peptic ulcer and gastrointestinal bleeding in the past 5 years.
* Patients have history of long-term (current) use of anticoagulants, spontaneous intracranial hemorrhage, and venous thromboembolism.
* Individuals have intracranial hemorrhage after surgery, or other active bleeding.
* Postoperative coagulation disorders (INR >1.5 or platelet counts < 100x10^9/L).
* Patients are allergic to Rivaroxaban.
* Pregnancy or breast-feeding women.
* Inability to give written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Venous thromboembolism | 6 months
  The occurrence of venous thromboembolism, including pulmonary embolism and venous thrombosis of the lower extremities.

SECONDARY OUTCOMES:
Fatal hemorrhage | 6 months
  Hemoglobin decreases by more than 20 g/L in 24 hours; Intracranial, intraspinal, intraocular, pericardial, retroperitoneal hemorrhage; other life-threatening hemorrhage.
Non-fatal hemorrhage | 6 months
  Wound hematomas, Ecchymosis, gastrointestinal bleeding, hemoptysis, hematuria, epistaxis; other non-fatal hemorrhage.

CONTACTS AND LOCATIONS:
Overall Officials: Guanglong Huang, M.D., Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (8):
- China (8):
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Fujian provincial hospital, Fuzhou, Fujian
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - The First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Longgang Central Hospital of Shenzhen, Shenzhen, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Hainan general hospital, Haikou, Hainan
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heit JA, Silverstein MD, Mohr DN, Petterson TM, O'Fallon WM, Melton LJ 3rd. Risk factors for deep vein thrombosis and pulmonary embolism: a population-based case-control study. Arch Intern Med. 2000 Mar 27;160(6):809-15. doi: 10.1001/archinte.160.6.809. PMID 10737280
- [Background] Khorana AA, Francis CW, Culakova E, Kuderer NM, Lyman GH. Thromboembolism is a leading cause of death in cancer patients receiving outpatient chemotherapy. J Thromb Haemost. 2007 Mar;5(3):632-4. doi: 10.1111/j.1538-7836.2007.02374.x. No abstract available. PMID 17319909
- [Background] Horsted F, West J, Grainge MJ. Risk of venous thromboembolism in patients with cancer: a systematic review and meta-analysis. PLoS Med. 2012;9(7):e1001275. doi: 10.1371/journal.pmed.1001275. Epub 2012 Jul 31. PMID 22859911
- [Background] Gerber DE, Grossman SA, Streiff MB. Management of venous thromboembolism in patients with primary and metastatic brain tumors. J Clin Oncol. 2006 Mar 10;24(8):1310-8. doi: 10.1200/JCO.2005.04.6656. PMID 16525187
- [Background] Knovich MA, Lesser GJ. The management of thromboembolic disease in patients with central nervous system malignancies. Curr Treat Options Oncol. 2004 Dec;5(6):511-7. doi: 10.1007/s11864-004-0039-x. PMID 15509484
- [Background] Tabori U, Beni-Adani L, Dvir R, Burstein Y, Feldman Z, Pessach I, Rechavi G, Constantini S, Toren A. Risk of venous thromboembolism in pediatric patients with brain tumors. Pediatr Blood Cancer. 2004 Nov;43(6):633-6. doi: 10.1002/pbc.20149. PMID 15390288
- [Background] Brandes AA, Scelzi E, Salmistraro G, Ermani M, Carollo C, Berti F, Zampieri P, Baiocchi C, Fiorentino MV. Incidence of risk of thromboembolism during treatment high-grade gliomas: a prospective study. Eur J Cancer. 1997 Sep;33(10):1592-6. doi: 10.1016/s0959-8049(97)00167-6. PMID 9389920
- [Background] Simanek R, Vormittag R, Hassler M, Roessler K, Schwarz M, Zielinski C, Pabinger I, Marosi C. Venous thromboembolism and survival in patients with high-grade glioma. Neuro Oncol. 2007 Apr;9(2):89-95. doi: 10.1215/15228517-2006-035. Epub 2007 Feb 27. PMID 17327573
- [Background] Dhami MS, Bona RD, Calogero JA, Hellman RM. Venous thromboembolism and high grade gliomas. Thromb Haemost. 1993 Sep 1;70(3):393-6. PMID 8259536
- [Background] Collins A, Sundararajan V, Brand CA, Moore G, Lethborg C, Gold M, Murphy MA, Bohensky MA, Philip J. Clinical presentation and patterns of care for short-term survivors of malignant glioma. J Neurooncol. 2014 Sep;119(2):333-41. doi: 10.1007/s11060-014-1483-5. Epub 2014 Jun 3. PMID 24889839
- [Background] Tucha O, Smely C, Preier M, Lange KW. Cognitive deficits before treatment among patients with brain tumors. Neurosurgery. 2000 Aug;47(2):324-33; discussion 333-4. doi: 10.1097/00006123-200008000-00011. PMID 10942005
- [Background] Chaichana KL, Pendleton C, Jackson C, Martinez-Gutierrez JC, Diaz-Stransky A, Aguayo J, Olivi A, Weingart J, Gallia G, Lim M, Brem H, Quinones-Hinojosa A. Deep venous thrombosis and pulmonary embolisms in adult patients undergoing craniotomy for brain tumors. Neurol Res. 2013 Mar;35(2):206-11. doi: 10.1179/1743132812Y.0000000126. Epub 2012 Dec 13. PMID 23336127
- [Background] Jenkins EO, Schiff D, Mackman N, Key NS. Venous thromboembolism in malignant gliomas. J Thromb Haemost. 2010 Feb;8(2):221-7. doi: 10.1111/j.1538-7836.2009.03690.x. Epub 2009 Nov 13. PMID 19912518
- [Background] Misch M, Czabanka M, Dengler J, Stoffels M, Auf G, Vajkoczy P, Stockhammer F. D-dimer elevation and paresis predict thromboembolic events during bevacizumab therapy for recurrent malignant glioma. Anticancer Res. 2013 May;33(5):2093-8. PMID 23645760
- [Background] Perry JR, Julian JA, Laperriere NJ, Geerts W, Agnelli G, Rogers LR, Malkin MG, Sawaya R, Baker R, Falanga A, Parpia S, Finch T, Levine MN. PRODIGE: a randomized placebo-controlled trial of dalteparin low-molecular-weight heparin thromboprophylaxis in patients with newly diagnosed malignant glioma. J Thromb Haemost. 2010 Sep;8(9):1959-65. doi: 10.1111/j.1538-7836.2010.03973.x. PMID 20598077
- [Background] Mohamed MFH, ElShafei MN, Ahmed MB, Abdalla LO, Ahmed I, Elzouki AN, Danjuma MI. The Net Clinical Benefit of Rivaroxaban Compared to Low-Molecular-Weight Heparin in the Treatment of Cancer-Associated Thrombosis: Systematic Review and Meta-Analysis. Clin Appl Thromb Hemost. 2021 Jan-Dec;27:1076029620940046. doi: 10.1177/1076029620940046. PMID 33651658
- [Background] Young AM, Marshall A, Thirlwall J, Chapman O, Lokare A, Hill C, Hale D, Dunn JA, Lyman GH, Hutchinson C, MacCallum P, Kakkar A, Hobbs FDR, Petrou S, Dale J, Poole CJ, Maraveyas A, Levine M. Comparison of an Oral Factor Xa Inhibitor With Low Molecular Weight Heparin in Patients With Cancer With Venous Thromboembolism: Results of a Randomized Trial (SELECT-D). J Clin Oncol. 2018 Jul 10;36(20):2017-2023. doi: 10.1200/JCO.2018.78.8034. Epub 2018 May 10. PMID 29746227